CLINICAL TRIAL: NCT01131169
Title: A Trial of Busulfan, Melphalan, Fludarabine and T-Cell Depleted Allogeneic Hematopoietic Stem Cell Transplantation Followed by Post Transplantation Donor Lymphocyte Infusions for Patients With Relapsed or High-Risk Multiple Myeloma
Brief Title: Busulfan, Melphalan, Fludarabine and T-Cell Depleted Allogeneic Hematopoietic Stem Cell Transplantation Followed by Post Transplantation Donor Lymphocyte Infusions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Otsuka America Pharmaceutical (Industry); Ludwig Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-051
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2019-06

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Busulfan; Melphalan; Fludarabine; T-Cell; Stem Cell Transplantation; 10-051
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Busulfan; Melphalan; fludarabine

ARMS (2):
- relapsed multiple myeloma (Experimental): This is a two arm phase II trial to assess the progression-free and overall survival as well as the safety and efficacy of allogeneic hematopoietic stem cell transplantation using a preparative regimen with busulfan, melphalan, fludarabine, and anti-thymocyte globulin (ATG), and a T cell depleted stem cell transplant from a histocompatible related or unrelated donor in patients with relapsed or high-risk multiple myeloma.
  Interventions: Drug: busulfan, melphalan and fludarabine
- high-risk multiple myeloma (Experimental): This is a two arm phase II trial to assess the progression-free and overall survival as well as the safety and efficacy of allogeneic hematopoietic stem cell transplantation using a preparative regimen with busulfan, melphalan, fludarabine, and anti-thymocyte globulin (ATG), and a T cell depleted stem cell transplant from a histocompatible related or unrelated donor in patients with relapsed or high-risk multiple myeloma.
  Interventions: Drug: busulfan, melphalan and fludarabine

INTERVENTIONS:
Drug: busulfan, melphalan and fludarabine — Patients will be cytoreduced with IV busulfan, melphalan and fludarabine. Busulfan will be administered at a dose of 0.8mg/Kg q6hrs for 10 doses on days -9, -8, -7. Doses for busulfan should be adjusted according to pharmacokinetic studies. Melphalan will be administered at a dose of 70 mg/m2/day for 2 days on days -7, -6. Fludarabine will be administered at a dose of 25 mg/m2/day for 5 days on days -6, -5, -4, -3, -2. Patients will also receive rabbit anti-thymocyte globulin (ATG) to prevent immune mediated graft rejection. The ATG will be administered at a dose of 2.5 mg/Kg/day IV on days -3 and -2. Doses for busulfan, melphalan and ATG should be adjusted if patient is > 125% ideal body weight and should be calculated on adjusted ideal body weight.
  Other Names: Doses of fludarabine should be reduced to 80% of dose for measured creatinine; clearance of 40-70ml/min. Day - 1 will be a day of rest before receiving the; T-cell depleted stem cell product on day 0. The preferred stem cell product; will be peripheral blood stem cells but if the donor is unable or unwilling to; donate peripheral blood stem cells, bone marrow will be used as the stem cell; source. Patients will receive post-transplant G-CSF starting on day +7.
  Arms: relapsed multiple myeloma
Drug: busulfan, melphalan and fludarabine — Patients will be cytoreduced with IV busulfan, melphalan and fludarabine. Busulfan will be administered at a dose of 0.8mg/Kg q6hrs for 10 doses on days -9, -8, -7. Doses for busulfan should be adjusted according to pharmacokinetic studies. Melphalan will be administered at a dose of 70 mg/m2/day for 2 days on days -7, -6. Fludarabine will be administered at a dose of 25 mg/m2/day for 5 days on days -6, -5, -4, -3, -2. Patients will also receive rabbit anti-thymocyte globulin (ATG) to prevent immune mediated graft rejection. The ATG will be administered at a dose of 2.5 mg/Kg/day IV on days -3 and -2. Doses for busulfan, melphalan and ATG should be adjusted if patient is > 125% ideal body weight and should be calculated on adjusted ideal body weight.
  Other Names: Doses of fludarabine should be reduced to 80% of dose for measured creatinine; clearance of 40-70ml/min. Day - 1 will be a day of rest before receiving the; T-cell depleted stem cell product on day 0. The preferred stem cell product; will be peripheral blood stem cells but if the donor is unable or unwilling; to donate peripheral blood stem cells, bone marrow will be used as the stem cell; source. Patients will receive post-transplant G-CSF starting on day +7.
  Arms: high-risk multiple myeloma

SUMMARY:
The patients are being offered a stem cell transplant. Stem cells are very early blood cells. They have not yet matured to become red or white blood cells or platelets. They have already received the standard treatment of chemotherapy and an autologous stem cell transplant. An autologous stem cell transplant is when the patient receives their infusion of their own cells. Thi will give the patient a better chance of curing the disease, this protocol includes an infusion of stem cells from the blood (or the bone marrow) of another person. This is called an allogeneic stem cell transplant. The stem cells will begin to grow in the bone marrow and produce new blood cells.

Allogeneic stem cell transplants can cause a condition called graft-versus-host disease or GVHD. In GVHD, a kind of white blood cell from the donor (graft) begins to attack the body (host). That blood cell is called a T-cell. It is a cell that normally helps to protects against things like bacteria and viruses. In this case, the donor's T-cells see the body as foreign in the same way they would see bacteria as foreign. GVHD can be fatal. In order to lower the chance that the patient will get GVHD this protocol treatment will remove the T-cells from the donor's cells. This is called T-cell depletion. The T cells are removed by a system called "Clinimacs". This method is still being evaluated through clinical trials and not been approved by the Federal Drug Administration (FDA) at this time.

Before the transplant, the physician will treat the bone marrow to get rid of the cancer. The physician uses three chemotherapy drugs plus ATG. The chemotherapy drugs (Busulfan, Melphalan and Fludarabine) kills the cancer. ATG gets rid of any of the patients T cells that survive the chemotherapy. This ensures that the donor stem cells are not rejected. The patient will also receive additional white blood cells called lymphocytes from the donor. This is called a donor lymphocyte infusion or DLI. These additional infusions will help cause a graft-versus-myeloma effect and can help the donor stem cells grow.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have multiple myeloma that has either relapsed or has high risk cytogenetics.
* Patients with relapsed multiple myeloma following autologous stem cell transplantation must have achieved at least partial response following additional chemotherapy (cohort 1):
* Patients are eligible if relapse occurs with complex/high-risk cytogenetics or occurs with normal cytogenetics but within 15 months following the autologous transplant.
* Patients with high risk cytogenetics at diagnosis must have achieved at least very good partial response following autologous stem cell transplantation (cohort 2):

  * Patients must have complex karyotype, 1q25, del17p, t4;14 and/or t14;16 by FISH and/or del13 by karyotyping.

DONOR: Patients must have a healthy HLA matched or mismatched related or unrelated donor who is willing to receive G-CSF injections and undergo apheresis for PBSC collection, or undergo a marrow harvesting procedure.

1. HLA-matched related and unrelated donors Patients who have an HLA-matched related or unrelated donor are eligible for entry on this protocol. This will include a healthy donor who is genotypically matched at all A, B, C, DRB1 and DQB1 locus, loci, as tested by DNA analysis.
2. HLA- mismatched related and unrelated donors Patients who do not have an HLA-matched donor but have a related or unrelated donor who have one antigen or one allele mismatch at the HLA A, B, C, DRB1 or DQB1 loci; or who have two mismatches, at HLA-DQB1 and at one other locus, will be eligible for entry on this protocol.

The following inclusion criteria are also required:

* Patients should be ≥ 21, < 73 years old.
* Patients may be of either gender or any ethnic background.
* Patients must have a Karnofsky (adult) or Performance Status ≥ 70%
* Patients must have adequate organ function measured by:

Cardiac: asymptomatic or if symptomatic then LVEF at rest must be ≥ 50% and must improve with exercise. Hepatic: < 3x ULN ALT and ≤ 1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia.

Renal: serum creatinine <1.2 mg/dl or if serum creatinine is outside the normal range, then CrCl > 40 ml/min (measured or calculated/estimated) with dose adjustment of Fludarabine for <70ml/min.

Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted (corrected for hemoglobin)

* Each patient must be willing to participate as a research subject and must sign an informed consent form.

Exclusion Criteria:

* Patients achieving < Partial Response following preceding chemotherapy (cohort 1) or < Very Good Partial Response following autologous stem cell transplantation (cohort 2).
* Patients with Plasma Cell Leukemia.
* Female patients who are pregnant or breast-feeding
* Active viral, bacterial or fungal infection
* Patient seropositive for HIV-I/II; HTLV -I/II
* Patients who have undergone prior allogeneic hematopoietic stem cell transplantation.
* Patients who have had a previous malignancy that is not in remission.
* Patients with known hypersensitivity to mouse proteins (murine antibodies in ISOLEX) if receiving SBA-E- bone marrow, or chicken egg products.

Ages: 21 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Tyler EM, Jungbluth AA, O'Reilly RJ, Koehne G. WT1-specific T-cell responses in high-risk multiple myeloma patients undergoing allogeneic T cell-depleted hematopoietic stem cell transplantation and donor lymphocyte infusions. Blood. 2013 Jan 10;121(2):308-17. doi: 10.1182/blood-2012-06-435040. Epub 2012 Nov 16. PMID 23160468
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Relapsed Multiple Myeloma | High-risk Multiple Myeloma
Started | 47 | 19
Completed | 47 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relapsed Multiple Myeloma | High-risk Multiple Myeloma | Total
Number analyzed (Participants) | 47 | 19 | 66
Age, Continuous [Mean (Full Range); unit: years] | 55.3 [37 to 66] | 49.5 [38 to 62] | 54 [37 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 35 | 14 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 42 | 17 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 34 | 17 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 19 | 65
  Turkey | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Relapsed Multiple Myeloma With Progression-free (PFS)
Time Frame: 2 years
Population: This objective only applies to Arm I: Participants with Relapsed Multiple Myeloma
Measure: Number (95% Confidence Interval); unit: Proportion of participants PFS
Arm/Group | Relapsed Multiple Myeloma | High-risk Multiple Myeloma
Number analyzed (Participants) | 47 | 0
Proportion of participants PFS | 0.31 [0.19 to 0.5] |

2. Secondary Outcome: Proportion of Participants With Relapsed Multiple Myeloma Alive at 2 Years
Time Frame: 2 years
Population: This objective is only for participants with relapsed multiple myeloma.
Measure: Number (95% Confidence Interval); unit: Proportion of pts alive at 2 years
Arm/Group | Relapsed Multiple Myeloma | High-risk Multiple Myeloma
Number analyzed (Participants) | 44 | 0
Proportion of pts alive at 2 years | 0.54 [0.41 to 0.72] |

3. Secondary Outcome: Number of Participants Who Relapse That Are Restored to Remission (CR)
Description: To compute the current multiple myeloma free survival curve in order to account for patients who relapse and are restored to remission through DLI.
Time Frame: 3 years
Population: This group consists of participants with residual disease either because they did not reach CR from salvage and transplant conditioning or because they were given this dose at the time of progression
Measure: Count of Participants; unit: Participants
Arm/Group | Relapsed Multiple Myeloma
Number analyzed (Participants) | 18
Participants
  Restored to CR, did not develop GVHD | 4
  Were not restored to CR, did not develop GVHD | 14

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 years
Arm/Group | Relapsed Multiple Myeloma | High-risk Multiple Myeloma
All-Cause Mortality (participants affected / at risk) | 17/47 | 9/19
Serious Adverse Events (participants affected / at risk) | 29/47 | 11/19
Other Adverse Events (participants affected / at risk) | 47/47 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relapsed Multiple Myeloma (N=47) | High-risk Multiple Myeloma (N=19)
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 2 | 0
Confusion (Psychiatric disorders) | 1 | 0
Creatinine increased (Investigations) | 0 | 1
Death NOS (General disorders) | 9 | 2
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 4
Dizziness (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Fatigue (General disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Fever (General disorders) | 4 | 0
Gen disorders & admin site conditions Other, spec (General disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Inf norm ANC/gr1/2 neut-Pneumonia(lung) (Infections and infestations) | 1 | 2
Infection, other (Infections and infestations) | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 17 | 4
Lethargy (Nervous system disorders) | 1 | 0
Lung infection (Infections and infestations) | 7 | 0
Nausea (Gastrointestinal disorders) | 6 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Neurology - Other (specify) (Nervous system disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Platelet count decreased (Investigations) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 4 | 0
Sinusitis (Infections and infestations) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relapsed Multiple Myeloma (N=47) | High-risk Multiple Myeloma (N=19)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0
Hypotension (Vascular disorders) | 3 | 0
Pain (General disorders) | 3 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 | 0
Fatigue (General disorders) | 4 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 3
Weight loss (Investigations) | 5 | 5
Mucositis oral (Gastrointestinal disorders) | 5 | 6
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 6 | 4
Anorexia (Metabolism and nutrition disorders) | 6 | 6
Activated partial thromboplastin time prolonged (Investigations) | 7 | 3
Alanine aminotransferase increased (Investigations) | 33 | 12
Alkaline phosphatase increased (Investigations) | 22 | 7
Aspartate aminotransferase increased (Investigations) | 30 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT01131169/Prot_SAP_000.pdf